CLINICAL TRIAL: NCT06004973
Title: Usability of STAR Particles in Healthy Volunteers: A Pilot Study
Brief Title: Aldena STAR Particles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Eric Felner, Professor of Medicine, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00005486; 2024P008520 (Other: Emory IRB)
Record Dates: First submitted 2023-06-18; First posted 2023-08-22 (Actual); Results first posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: STAR particles; Skin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- STAR Particles application (Experimental): Participants will receive the 8 interventions (different application pressures) plus the control (Site and treatment will not be randomly assigned on the arm) by the investigator.
  Interventions: Device: STAR Particles
- Control Application (Other): Participants 1 to 10 will receive one control application on the volar side of one forearm.
  Participants 11 to 20 will receive one control application on the opposite forearm and on the contralateral side of the face.
  Interventions: Device: Gel without STAR Particles

INTERVENTIONS:
Device: STAR Particles — A 1.5-gram dose of STAR particles (10% concentration in aloe vera ointment) will be applied to the eight application sites (forearm and hand). Two rubbing cycles (30 and 60 cycles at a minimum of 1 cycle/second) and three pressures (40, 60, and 80 kPa) will be evaluated
  Arms: STAR Particles application
Device: Gel without STAR Particles — A 100mg dose of the gel without STAR particles is applied to the control site (the forearm for all participants and, additionally, the face for participants 11-20).
  Other Names: Control
  Arms: Control Application

SUMMARY:
The objective of this study is to find out the best method of applying STAR particles to the skin. STAR particles are very small particles with microneedles on the surface that can increase and create small punctures in the skin.

The small punctures should allow for different topical medications to work more effectively. This is important to understand the potential use of STAR particles in future topical medications. This study will not use any medication with active ingredients.

The study will include healthy adult participants. The first visit will be to collect medical information and assess eligibility in the study. The second visit will have the application of STAR particles on different areas of the arm, hand, and face with different pressures to determine what the most effective method of application is. The skin will be evaluated after the application, and surveys will be collected on the tolerability of the application.

DETAILED DESCRIPTION:
The goal of this study is to identify the most efficacious pressure of administration and the minimum number of rubbing cycles necessary to perforate the stratum corneum (the outermost layer of the skin).

Many medical conditions are treated through the topical application of a therapeutic compound formulated into a gel, cream, ointment, or lotion (e.g., eczema, psoriasis, actinic keratosis, cutaneous warts). This is especially true in dermatology, in which the skin is often the primary site of action. Topicals (i.e., drugs applied to the skin's surface) allow patients to easily self-apply these therapies without the need for painful or difficult-to-use medical technologies (e.g., hypodermic needles) or the risks associated with systemic exposure to a drug (e.g., oral, intravenous, or intramuscular administration).

Despite the advantages associated with topical delivery, the skin serves as a barrier to the transport of most external compounds. There are several techniques to overcome the skin barrier. Several studies have been conducted to increase skin permeability using various methods, including chemical, biochemical, and physical approaches. However, chemical and biochemical methods do not appear to be broadly useful for the delivery of large molecule therapeutics (e.g., peptides, proteins, genetic material) across the skin. STAR particles are millimeter-scale particles with micron-scale projections made of biocompatible materials that painlessly disrupt the stratum corneum. As STAR particles are rubbed on the skin, their microscopic projections create micron-scale pores in the stratum corneum to increase skin permeability to topical compounds independent of physicochemical properties. After the arms of the STAR particle puncture the skin, the elastic forces of the skin push the particles out. The first 10 participants will receive the 8 interventions (different application pressures) plus the control (Site and treatment will not be randomly assigned to the arm) by the investigator. In addition, two applications of STAR particles will be applied to one of the hands. After these participants have completed the study, an interim analysis will be performed. At this point, a decision will be made by the investigator to determine if changes in STAR particle administration will be implemented for the next 10 participants.

ELIGIBILITY:
Inclusion Criteria:

* Adult, 18 - 39 years of age
* In good general health as determined by a medical history
* Willing and able to provide informed consent and follow all study requirements
* Not pregnant and does not desire to become pregnant in the subsequent two months

Exclusion Criteria:

* Has a known allergy or sensitivity to aloe vera or alumina
* Has any skin disorders or skin allergies
* Has any medical condition that may affect skin or skin sensation
* Has abnormal (e.g., tattooed) skin at forearms
* Has known neurological condition affecting sensory function or perception of pain
* Has inflammatory bowel disease
* Has applied skin ointment or cream to forearms in the previous 24 hours
* Has a major congenital or chromosomal abnormality known to affect the skin
* Has taken pain medication in the last 24 hours
* Is currently participating in another interventional clinical trial
* Has previously participated in a STAR particle interventional clinical trial
* Is pregnant or wishing to be pregnant
* Has any condition (social or medical), which in the opinion of the investigator would make study participation unsafe, would interfere with adherence to the clinical study requirements, or would complicate data interpretation

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric I Felner, MD, MSCR, Principal Investigator — Emory University
Locations (1):
- Emory Children's Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in Atlanta, Georgia, USA. Participant enrollment began February 7, 2024, and all follow-up was complete by December 7, 2024.
Pre-assignment Details: This was an ADAPTIVE STUDY DESIGN so that after reviewing the data collected from the first 10 participants (Part 1), conditions were altered so that the ideal conditions (cycles and pressure application) discovered from Part 1 (first 10 participants) would be used for the next 10 participants (11 - 20) in Part 2 of the study. In Part 2, each subject had STARs applied to the right head/face and the right forearm, and a control was applied to the left head/face and the left forearm.
Groups:
- STAR Particles Part 1: Participants will receive the 8 interventions (different application pressures) plus the control (Site and treatment will not be randomly assigned on the arm) by the investigator.
  STAR Particles: A 1.5-gram dose of STAR particles (10% concentration in aloe vera ointment) will be applied to the eight application sites (forearm and hand) and 100 mg of aloe vera will be applied to the control site on one of the forearms. Two rubbing cycles (20 and 30 cycles at 1 cycle/second) and three pressures (40, 60, and 80 kPa) will be evaluated.
- STAR Particle Part 2: Participants in Part 2 will receive the STAR particle applications (one on the forearm and one on the side of the face) and one control application on the other forearm and on the other side of the face.
  STAR Particles: A 1.5-gram dose of STAR particles (10% concentration in aloe vera ointment) will be applied to the eight application sites (forearm and hand), and 100 mg of aloe vera will be applied to the control site on one of the forearms. Two rubbing cycles (60 cycles at 1 cycle/second and 80 kPa) will be evaluated.
Period: Part 1 (Participants 1-10)
Arm/Group | STAR Particles Part 1 | STAR Particle Part 2
Started (The first 10 participants received eight applications (three on each forearm and two to one hand) of STAR particles and one control application on the volar side of one of the forearms for a total of nine applications to the forearms.) | 10 | 0
Site 1: STAR Particles on forearm, 60 rubbing cycles/min at 40 kPa | 10 | 0
Site 2: STAR Particles on forearm, 60 rubbing cycles/min at 60 kPa | 10 | 0
Site 3: STAR Particles on forearm, 60 rubbing cycles/min at 80 kPa | 10 | 0
Site 4: Control Gel without STAR Particles on forearm, 30 rubbing cycles/min, 60 kPa | 10 | 0
Site 5: STAR Particles on forearm, 30 rubbing cycles/min at 80 kPa | 10 | 0
Site 6: STAR Particles on forearm, 30 rubbing cycles/min at 60 kPa | 10 | 0
Site 7: STAR Particles on forearm, 30 rubbing cycles/min at 40 kPa | 10 | 0
Site 8: STAR Particles on palm of hand, 30 rubbing cycles/min at 60 kPa | 10 | 0
Site 9: STAR Particles on dorsum of hand, 30 rubbing cycles/min at 60 kPa | 10 | 0
Completed | 10 | 0
Not Completed | 0 | 0
Period: Part 2 (Participants 11-20)
Arm/Group | STAR Particles Part 1 | STAR Particle Part 2
Started (Participants 11-20: Each participant had the STAR applications on the forearm and on the side of the face and one control application on the other forearm, and on the other side of the face.) | 0 | 10
STAR Particles on the Right Forearm | 0 | 10
STAR Particles on the Right Face (Forehead) | 0 | 10
Control Gel Application without STAR Particles on the Left Arm | 0 | 10
Control Gel Application without STAR Particles on the Left head (Forehead) | 0 | 10
Completed | 0 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Twenty participants enrolled: Participants 1-10 (9 application sites each) were used to determine ideal pressure & TEWL. Participants 11-20 had pain and sensation assessed at the forearms and face at the pressure and cycle levels previously chosen from the first 10 enrolled participants.
Groups:
- STAR Particles Part 1: Part 1 (Participants 1-10): Each participant received eight interventions (different application pressures) plus one control. Sites and treatments were not randomly assigned to arms; the investigator administered all applications.
- STAR Particles Part 2: Part 2 (Participants 11-20): Conditions were adjusted based on the findings from Part 1, so that the optimal cycles and pressure application identified earlier could be applied. Each participant received STAR applications to the right head/face and right forearm, and a control application to the left head/face and left forearm.
- Total: Total of all reporting groups
Arm/Group | STAR Particles Part 1 | STAR Particles Part 2 | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.71 (5.45) | 25.50 (5.47) | 25.55 (5.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 2 | 5 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 9 | 5 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 5 | 3 | 8
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 5 | 5
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Transepidermal Water Loss (TEWL)
Description: Trans-epidermal water loss (TEWL) measurement (only for the first 10 participants 1-10) before and after application of STAR particles [(T0 (before), T20 (after), T30 (after)].
Time Frame: Before application, 20 minutes after application, and 30 minutes after application
Population: Participants 1-10, who had TEWL measurements.
Measure: Mean (Standard Deviation); unit: g/m^2/hr
Groups:
- Site 1: STAR Particles on Right Forearm, 60 Rubbing Cycles/Min at 40 kPa Pressure: Site 1: STAR Particles on Right forearm, 60 Rubbing Cycles/Min at 40 kPa pressure
  Participants 1-10 will receive the 8 interventions (different application pressures) plus the control (Site and treatment will not be randomly assigned to an arm) from the investigator.
  STAR Particles: A 1.5-gram dose of STAR particles (10% concentration in aloe vera ointment) will be applied to the eight application sites (forearm and hand), and 100 mg of aloe vera will be applied to the control site on one of the forearms. Two rubbing cycles (20 and 30 cycles at 1 cycle/second) and three pressures (40, 60, and 80 kPa) will be evaluated.
- Site 2 -STAR Particles on Right Forearm, 60 Rubbing Cycles/Min at 60 kPa Pressure: Site 2 -STAR Particles on Right forearm, 60 Rubbing Cycles/min at 60 kPa pressure
  Participants 1-10 will receive the 8 interventions (different application pressures) plus the control (Site and treatment will not be randomly assigned to an arm) from the investigator.
  STAR Particles: A 1.5-gram dose of STAR particles (10% concentration in aloe vera ointment) will be applied to the eight application sites (forearm and hand), and 100 mg of aloe vera will be applied to the control site on one of the forearms. Two rubbing cycles (20 and 30 cycles at 1 cycle/second) and three pressures (40, 60, and 80 kPa) will be evaluated.
- Site 3: STAR Particles on Right Forearm, 60 Rubbing Cycles/Min at 80 kPa: Site 3: STAR particles on Right forearm, 60 Rubbing Cycles/Min at 80 kPa
  Participants 1-10 will receive the 8 interventions (different application pressures) plus the control (Site and treatment will not be randomly assigned to an arm) from the investigator.
  STAR Particles: A 1.5-gram dose of STAR particles (10% concentration in aloe vera ointment) will be applied to the eight application sites (forearm and hand), and 100 mg of aloe vera will be applied to the control site on one of the forearms. Two rubbing cycles (20 and 30 cycles at 1 cycle/second) and three pressures (40, 60, and 80 kPa) will be evaluated.
- Site 4: Control Gel on Left Forearm, 30 Rubbing Cycles/Min at 60 kPa Pressure: Site 4: Control Gel: Left forearm, 30 Rubbing Cycles/Min at 60 kPa pressure
  Participants 1-10 will receive the 8 interventions (different application pressures) plus the control (Site and treatment will not be randomly assigned to an arm) from the investigator.
  STAR Particles: A 1.5-gram dose of STAR particles (10% concentration in aloe vera ointment) will be applied to the eight application sites (forearm and hand), and 100 mg of aloe vera will be applied to the control site on one of the forearms. Two rubbing cycles (20 and 30 cycles at 1 cycle/second) and three pressures (40, 60, and 80 kPa) will be evaluated.
- Site 5: STAR Particles on Left Forearm, 30 Rubbing Cycles/Min at 80 kPa Pressure: Site 5: STAR Particles on Left forearm, 30 Rubbing Cycles/Min at 80 kPa pressure
  Participants 1-10 will receive the 8 interventions (different application pressures) plus the control (Site and treatment will not be randomly assigned to an arm) from the investigator.
  STAR Particles: A 1.5-gram dose of STAR particles (10% concentration in aloe vera ointment) will be applied to the eight application sites (forearm and hand), and 100 mg of aloe vera will be applied to the control site on one of the forearms. Two rubbing cycles (20 and 30 cycles at 1 cycle/second) and three pressures (40, 60, and 80 kPa) will be evaluated.
- Site 6: STAR Particles on Left Forearm, 30 Rubbing Cycles/Min at 60 kPa Pressure: Site 6: STAR Particles on Left forearm, 30 Rubbing Cycles/Min at 60 kPa pressure
  Participants 1-10 will receive the 8 interventions (different application pressures) plus the control (Site and treatment will not be randomly assigned to an arm) from the investigator.
  STAR Particles: A 1.5-gram dose of STAR particles (10% concentration in aloe vera ointment) will be applied to the eight application sites (forearm and hand), and 100 mg of aloe vera will be applied to the control site on one of the forearms. Two rubbing cycles (20 and 30 cycles at 1 cycle/second) and three pressures (40, 60, and 80 kPa) will be evaluated.
- SITE 7: STAR Particles on Left Forearm, 30 Rubbing Cycles/Min at 40 kPa Pressure.: SITE 7: STAR particles on Left forearm, 30 Rubbing Cycles/Min at 40 kPa pressure.
  Participants 1-10 will receive the 8 interventions (different application pressures) plus the control (Site and treatment will not be randomly assigned to an arm) from the investigator.
  STAR Particles: A 1.5-gram dose of STAR particles (10% concentration in aloe vera ointment) will be applied to the eight application sites (forearm and hand), and 100 mg of aloe vera will be applied to the control site on one of the forearms. Two rubbing cycles (20 and 30 cycles at 1 cycle/second) and three pressures (40, 60, and 80 kPa) will be evaluated.
- Site 8: STAR Particles on the Palm of the Right Hand at 30 Rubbing Cycles/Minute at 60 kPa Pressure: Site 8: STAR Particles on the Palm of the Right Hand at 30 Rubbing Cycles/Minute at 60 kPa Pressure
  Participants 1-10 will receive the 8 interventions (different application pressures) plus the control (Site and treatment will not be randomly assigned to an arm) from the investigator.
  STAR Particles: A 1.5-gram dose of STAR particles (10% concentration in aloe vera ointment) will be applied to the eight application sites (forearm and hand), and 100 mg of aloe vera will be applied to the control site on one of the forearms. Two rubbing cycles (20 and 30 cycles at 1 cycle/second) and three pressures (40, 60, and 80 kPa) will be evaluated.
- Site 9: STAR Particles on the Dorsum of the Right Hand, 30 Rubbing Cycles/Min at 60 kPa Pressure: Site 9: STAR Particles on the dorsum of the Right Hand, 30 Rubbing Cycles/Min at 60 kPa pressure
  Participants 1-10 will receive the 8 interventions (different application pressures) plus the control (Site and treatment will not be randomly assigned to an arm) from the investigator.
  STAR Particles: A 1.5-gram dose of STAR particles (10% concentration in aloe vera ointment) will be applied to the eight application sites (forearm and hand), and 100 mg of aloe vera will be applied to the control site on one of the forearms. Two rubbing cycles (20 and 30 cycles at 1 cycle/second) and three pressures (40, 60, and 80 kPa) will be evaluated.
Arm/Group | Site 1: STAR Particles on Right Forearm, 60 Rubbing Cycles/Min at 40 kPa Pressure | Site 2 -STAR Particles on Right Forearm, 60 Rubbing Cycles/Min at 60 kPa Pressure | Site 3: STAR Particles on Right Forearm, 60 Rubbing Cycles/Min at 80 kPa | Site 4: Control Gel on Left Forearm, 30 Rubbing Cycles/Min at 60 kPa Pressure | Site 5: STAR Particles on Left Forearm, 30 Rubbing Cycles/Min at 80 kPa Pressure | Site 6: STAR Particles on Left Forearm, 30 Rubbing Cycles/Min at 60 kPa Pressure | SITE 7: STAR Particles on Left Forearm, 30 Rubbing Cycles/Min at 40 kPa Pressure. | Site 8: STAR Particles on the Palm of the Right Hand at 30 Rubbing Cycles/Minute at 60 kPa Pressure | Site 9: STAR Particles on the Dorsum of the Right Hand, 30 Rubbing Cycles/Min at 60 kPa Pressure
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
g/m^2/hr
  Before Application (T0) | 25.96 (15.20) | 20.44 (6.97) | 20.31 (7.89) | 23.82 (5.43) | 19.33 (2.96) | 21.44 (9.31) | 21.39 (5.64) | 560.15 (294.51) | 43.43 (11.21)
  20 minutes Post-Application (T20) | 20.94 (3.83) | 20.15 (2.71) | 20.31 (5.39) | 23.26 (5.81) | 23.29 (8.77) | 20.85 (5.22) | 20.12 (4.36) | 444.20 (218.29) | 41.33 (10.21)
  30 minutes Post - Application (T30) | 20.38 (3.11) | 18.88 (3.08) | 19.79 (4.84) | 22.38 (7.16) | 21.19 (4.95) | 20.42 (4.99) | 18.90 (4.21) | 290.45 (202.65) | 35.82 (8.33)

2. Secondary Outcome: Sensation After Application of STAR Particles (Part 2 Only)
Description: Measured using a Likert-type scale ranging from 0 to 5, where 0 = No Pain and 5 = Severe Pain. Higher scores indicate greater perceived sensation.
  Sensation was evaluated only among participants in the STAR Particles study, Part 2.
Time Frame: Immediately After STAR particles application
Population: Sensation was evaluated only among participants in Part 2 of the STAR Particles study (Participants 11-20).
Measure: Mean (Standard Deviation); unit: score on a Likert scale
Groups:
- STAR Particles (Part 2) on the Right Forearm, 60 Rubbing Cycles/Min at 80 KPa Pressure: STAR Particles on the Right Forearm, 60 Rubbing Cycles/Min at 80 KPa pressure.
  Participants will receive the 4 interventions (different application pressures).
  Participants received a 1.5-gram dose of STAR particles (10% concentration in aloe vera ointment) at the eight application sites (forearm and face)
- STAR Particles (Part 2) on the Right Face (Forehead), 60 Rubbing Cycles/Min at 80 KPa Pressure.: STAR Particles on the Right Face (Forehead), 60 Rubbing Cycles/Min at 80 KPa pressure.
  Participants will receive the 4 interventions (different application pressures)
  Participants received a 1.5-gram dose of STAR particles (10% concentration in aloe vera ointment) to the eight application sites (forearm and face).
- Part 2: Control Gel Application Without STAR Particles on the Left Forearm: Participants will receive one control application on the other forearm and on the other side of the face.
  100 mg of the gel without STAR particles will be applied to the control site on one of the forearms.
- Part 2: Control Gel Application Without STAR Particles on the Left Head (Forehead): Participants will receive the control application on the other side of their face.
  100 mg of gel without STAR particles will be applied to the control site on their face (forehead).
Arm/Group | STAR Particles (Part 2) on the Right Forearm, 60 Rubbing Cycles/Min at 80 KPa Pressure | STAR Particles (Part 2) on the Right Face (Forehead), 60 Rubbing Cycles/Min at 80 KPa Pressure. | Part 2: Control Gel Application Without STAR Particles on the Left Forearm | Part 2: Control Gel Application Without STAR Particles on the Left Head (Forehead)
Number analyzed (Participants) | 10 | 10 | 10 | 10
score on a Likert scale | 0.60 (0.43) | 0.60 (0.87) | 0.20 (0.43) | 0.10 (0)

3. Secondary Outcome: Evaluate Pain Using the Visual Analog Pain Scale (VAPS) After Application of the STAR Particles (Part 2 Only)
Description: The Visual Analog Pain Scale is a tool used to measure a person's pain intensity. It is a unidimensional scale, typically represented by a straight line often depicted as a 100 mm line with one end marked "no pain" (0) and the other marked "worst imaginable pain" (100). For this outcome, results will be reported as a percentage of the 100 mm VAPS scale, where 0% corresponds to no pain and 100% corresponds to the worst imaginable pain. A higher percentage indicates greater pain intensity.
  VAPS was evaluated only among participants in the STAR Particles study, Part 2.
Time Frame: Immediately After STAR particles application
Population: VAPS was evaluated only among participants in Part 2 of the STAR Particles study (Participants 11-20).
  For each participant, all application sites on the right arm were assessed, and the results were aggregated into a single value. Similarly, all application sites on the right side of the face were assessed and reported as a separate aggregated result.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- STAR Particles (Part 2) on the Right Forearm, 60 Rubbing Cycles/Min at 80 KPa Pressure: Participants will receive the STAR interventions (different application pressures)
  STAR Particles: A 1.5-gram dose of STAR particles (10% concentration in aloe vera ointment) will be applied to the application sites (forearm and face).
- STAR Particles (Part 2) on the Right Face (Forehead), 60 Rubbing Cycles/Min, at 80 kPa Pressure.: Participants will receive the STAR interventions (different application pressures)
  STAR Particles: A 1.5-gram dose of STAR particles (10% concentration in aloe vera ointment) will be applied to the eight application sites (forearm and face).
- Part 2: Control Gel Application Without STAR Particles on the Left Face (Forehead): Participants will receive the control application on the other side of the face.
  100 mg of gel without STAR particles will be applied to the control site on the face (forehead).
Arm/Group | STAR Particles (Part 2) on the Right Forearm, 60 Rubbing Cycles/Min at 80 KPa Pressure | STAR Particles (Part 2) on the Right Face (Forehead), 60 Rubbing Cycles/Min, at 80 kPa Pressure. | Part 2: Control Gel Application Without STAR Particles on the Left Forearm | Part 2: Control Gel Application Without STAR Particles on the Left Face (Forehead)
Number analyzed (Participants) | 10 | 10 | 10 | 10
score on a scale | 1.90 (1.64) | 2.70 (6.06) | 0.80 (0.87) | 0.10 (0)

4. Secondary Outcome: Number or Participants Who Reported Standard Adverse Event (AE)
Description: Number of participants during each period of participation who reported any adverse events after the removal of the STAR particles at any of the sites of application.
Time Frame: Up to 5 days after the STAR particles removal (for a total of 5 days)
Measure: Count of Participants; unit: Participants
Groups:
- STAR Particles (Part 1): Participants will receive the 8 interventions (different application pressures) plus the control (Site and treatment will not be randomly assigned on the arm) by the investigator.
  STAR Particles: A 1.5-gram dose of STAR particles (10% concentration in aloe vera ointment) will be applied to the eight application sites (forearm and hand), and 100 mg of aloe vera will be applied to the control site on one of the forearms. Two rubbing cycles (20 and 30 cycles at 1 cycle/second) and three pressures (40, 60, and 80 kPa) will be evaluated.
- STAR Particles (Part 2): Participants in Part 2 will receive the SRAR particle applications (one on the forearm and one on the side of the face of STAR particles, and one control application on the other forearm and on the other side of the face).
  STAR Particles: A 1.5-gram dose of STAR particles (10% concentration in aloe vera ointment) will be applied to the eight application sites (forearm and hand), and 100 mg of aloe vera will be applied to the control site on one of the forearms. Two rubbing cycles (60 cycles at 1 cycle/second and 80 kPa) will be evaluated.
Arm/Group | STAR Particles (Part 1) | STAR Particles (Part 2)
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

5. Other Pre Specified Outcome: Number of Participants Who Experience Adverse Events Due to Residual STAR Particles
Description: Participants will perform a visual inspection of the residual STAR particles after their removal and report any adverse events due to residual STAR particles up to 30 days after removal.
Time Frame: After STAR particles removal up to 30 days (for a total of 30 days)
Population: Because no serious adverse events (SAEs) occurred and the safety profile was consistent across all sites and study parts, safety data are reported in aggregate for all participants rather than by individual site or part. This approach was chosen to simplify reporting without compromising accuracy.
Measure: Count of Participants; unit: Participants
Groups:
- STAR Particles Part 1 and Part 2: Participants will receive the 8 interventions (different application pressures) plus the control (Site and treatment will not be randomly assigned on the arm) by the investigator.
  STAR Particles: A 1.5-gram dose of STAR particles (10% concentration in aloe vera ointment) will be applied to the eight application sites (forearm and hand) and 100 mg of aloe vera will be applied to the control site on one of the forearms. Two rubbing cycles (20 and 30 cycles at 1 cycle/second) and three pressures (40, 60, and 80 kPa) will be evaluated.
Arm/Group | STAR Particles Part 1 and Part 2
Number analyzed (Participants) | 20
Participants | 0

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected from the time of STAR particles application until 30 days after their removal, for a total observation period of 30 days.
Groups:
- STAR Particles Part 2: Participants will receive eight applications (one on the forearm and one on the side of the face of STAR particles, and one control application on the other forearm and on the other side of the face).STAR Particles: A 1.5-gram dose of
  STAR particles (10% concentration in aloe vera ointment) will be applied to the eight application sites (forearm and hand), and 100 mg of aloe vera will be applied to the control site on one of the forearms. Two rubbing cycles (60 cycles at 1 cycle/second and 80 kPa) will be evaluated.
Arm/Group | STAR Particles Part 1 | STAR Particles Part 2
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2024-04-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT06004973/Prot_000.pdf